CLINICAL TRIAL: NCT02332902
Title: Everolimus for Treatment of Disfiguring Cutaneous Lesions in Neurofibromatosis1- CRAD001CUS232T
Brief Title: Everolimus for Treatment of Disfiguring Cutaneous Lesions in Neurofibromatosis1 CRAD001CUS232T
Acronym: DCLNF1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Texas Neurofibromatosis Foundation (Unknown)
Responsible Party: Principal Investigator, Mary Kay Koenig, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-14-0758
Record Dates: First submitted 2014-12-12; First posted 2015-01-07 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Neurofibromatosis 1
Keywords: Neurofibroma; NF-1; Everolimus; mTOR inhibitor
MeSH Terms: conditions — Neurofibromatosis 1; Neurofibroma | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): This is a single arm intervention using Everolimus
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everyone in the study will receive Everolimus at a starting dose of 10 mg daily and will be adjusted up or down by 2.5 mg at 2 week intervals to attain a trough concentration of 5-15 ng/ml
  Other Names: Afinitor

SUMMARY:
This trial is evaluating the use of oral Everolimus to determine if there is a reduction in the size of the disfiguring cutaneous lesions in patients with Neurofibromatosis 1 over a 6 month period. The evaluation will be done by 3D photography measuring volume with the LIFEVIZ Micro system.

DETAILED DESCRIPTION:
Qualifying subjects will have a diagnosis of Neurofibromatosis 1 and have disfiguring cutaneous lesions that can be measured by photography. The subjects will have photographs of the target lesions,biopsies of the lesions,and safety blood laboratory tests at 3 time points (baseline, 3 months and 6 months which is end of treatment). Everolimus will be taken orally for 6 months. Subjects will visit the clinic monthly for an exam and adverse event evaluation. Laboratory testing will be done at these visits if determined necessary by the PI.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is at least 18 years of age at the time of enrollment
2. Informed consent
3. Compliance with trial requirements (photography, lab draws, medication schedules, and study visits)
4. Diagnosis of NF 1 and has cutaneous neurofibromas that are located in in a region amenable to photography
5. Females of child bearing potential must not be pregnant as confirmed by a negative pregnancy test (blood beta-hCG level) prior to study enrollment and must agree to use appropriate contraceptive methods for the duration of the trial
6. Patient must have adequate liver function as shown by, total bilirubin </= 2.0 mg/dL, ALT and AST </= 2.5 X ULN, INR </= 2

8. Patient must have adequate renal function, serum creatinine </= 1.5 X ULN 9. Patient must have adequate lipid profile, fasting serum cholesterol </= 300 mg/dL OR </= 7.75 mmol/L, fasting triglycerides </= X ULN

Exclusion Criteria:

1. Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of Everolimus (including chemotherapy, radiation therapy, antibody based therapy, etc.) 2. Known intolerance or hypersensitivity to Everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus) 3. Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral Everolimus 4. Uncontrolled diabetes mellitus despite adequate therapy 5. Patients who have any severe and /or uncontrolled medical conditions such as: unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction </= prior to start of Everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease, symptomatic congestive heart failure of New York Hear Association Class III or IV, known active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, or chronic hepatitis, known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air), active, bleeding diathesis, chronic treatment with corticosteroids, or other immunosuppressive agents, topical or inhaled corticosteroids are allowed, know history of HIV seropositivity, patients who have received live attenuated vaccines within 1 week of start of Everolimus. Patient would avoid close contact with others who have received live attenuated vaccines during the study, patients who have a history of primary malignancy, with the exceptions of mon-melanoma skin cancer, and carcinoma in situ of the cervix, uteri, or breast from which the patient has been disease free for >/- 3 years, patients with a history of non compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study, patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing, pregnant or nursing (lactating) women, women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing of study treatment. highly effective contraception methods,male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Koenig, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Result] Slopis JM, Arevalo O, Bell CS, Hebert AA, Northrup H, Riascos RF, Samuels JA, Smith KC, Tate P, Koenig MK. Treatment of Disfiguring Cutaneous Lesions in Neurofibromatosis-1 with Everolimus: A Phase II, Open-Label, Single-Arm Trial. Drugs R D. 2018 Dec;18(4):295-302. doi: 10.1007/s40268-018-0248-6. PMID 30284154

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 of the 24 enrolled participants withdrew consent immediately and did not receive study drug.
Groups:
- Intervention: This is a single arm intervention using Everolimus.
  Everyone in the study will receive Everolimus at a starting dose of 10 mg daily and will be adjusted up or down by 2.5 mg at 2-week intervals to attain a trough concentration of 5-15 ng/mL.
Period: Overall Study
Arm/Group | Intervention
Started | 24
Received Study Drug | 22
Completed | 17
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: 3D Photographic Measurement of Surface Volume of Cutaneous Neurofibroma Lesion
Description: Photographs of selected lesions to measure surface volume.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: mm^3
Arm/Group | Intervention
Number analyzed (Participants) | 17
mm^3
  Baseline | 32.54 [14.30 to 50.77]
  6 months | 33.93 [13.28 to 54.58]

2. Secondary Outcome: Number of Participants With Grade 3-4 Adverse Events
Description: Determination if orally administered Afinitor is safe in patients a indicated by lack of Grade 3-4 adverse events during the trial period.
Time Frame: 6 months
Population: The 2 participants who withdrew consent and did not receive study drug were not analyzed for adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 22
Participants | 0

3. Other Pre Specified Outcome: Determine How Orally Administered Everolimus Effects mTOR Signaling in NF-1 Tissues
Description: Quantification via immunohistochemical staining of PTEN, pS6, p4EBP-1, TSC2, mTOR, NF-1, pAKT, VEGF-A and IGF-IR expression in biopsied neurofibroma tissue samples.
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 22/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=22)
Stomatitis (Skin and subcutaneous tissue disorders) | 20 (20)
Upper Respiratory Infection/Cough/Sinus Infection/Pneumonia/Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Gastrointestinal (GI) Upset (Gastrointestinal disorders) | 9 (9)
Folliculitis/Impetigo/Rash/Itching (Skin and subcutaneous tissue disorders) | 9 (9)
Decreased Per Oral Intake/Weight loss (Gastrointestinal disorders) | 5 (5)
Headache (Nervous system disorders) | 3 (3)
Tooth Infection (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Fatigue (Nervous system disorders) | 3 (3)
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 2 (2)
Vaginitis (Infections and infestations) | 2 (2)
Thrush (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bladder Leakage (Renal and urinary disorders) | 1 (1)
Pheochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ingrown Toenail (Skin and subcutaneous tissue disorders) | 1 (1)
Nose Bleed (Vascular disorders) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1)
Left Side Numbness (Nervous system disorders) | 1 (1)
Biopsy Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Foggy Hearing (Ear and labyrinth disorders) | 1 (1)
Ammenorrhea (Reproductive system and breast disorders) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes